CLINICAL TRIAL: NCT05968092
Title: Role of US vs X Ray in Detection of Pediatric Elbow Fractures.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Mosad Shenouda, Resident doctor, Assiut University
Other Study IDs: US and X Ray in elbow
Record Dates: First submitted 2023-07-07; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Elbow Fractures
MeSH Terms: conditions — Elbow Fractures

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this prospective study is to evaluate and compare the accuracy of elbow ultrasonography with X Ray radiography for the diagnosis of elbow fractures in children following trauma in order to detect the validity of US in diagnosis of fractures as a dependent tool.

DETAILED DESCRIPTION:
Acute bone fractures in children are common and account for 10-25% of total injuries in early ages with considerable effects on activity restriction and subsequent high socioeconomical impact. In these cases, the elbow is a common site of pediatric fractures (account for up to 15% of all fractures) referring to the emergency department, and diagnostic testing with X-ray, including standard 2-way anteroposterior and lateral views, are required primarily for the evaluation of elbow injuries. In the setting of elbow trauma, the posterior fat pad sign on lateral radiographs is highly sensitive for fracture . However, radiological assessment of the elbow may be challenging in early ages due to the non-ossifed epiphysis and often non-exact two- plane radiographs in uncooperative children. Because of the higher sensitivity of growing bones to ionizing radiation, and dose-dependent radiation exposure is both CT scans and X-ray, every imaging should be minimized in children. Therefore, alternative imaging methods, such as US, have become a current issue to reduce exposure to radiation . Ultrasound is radiation-free, it is a real-time bedside assessment, it can be immediately performed and is easily accessible, and it is fast and reliable ,Ultrasonography can detect cortical disruption and irregularity, which directly indicates fractures. However, an elevated posterior fat pad can be easily identified by US, indirectly indicates intracapsular fractures . Ultrasonography is superior to radiography in detecting posterior fat pad elevation. Elbow joint effusion is a classic finding after trauma.

It is not always associated with a cortical fracture, whereas lipohaemarthrosis, corresponding to the presence of blood and lipid material in the posterior fat pad, indicates an intraarticular elbow fracture, too.

Lipohemarthrosis, as well as an elevated posterior fat pad, can easily be identifed on ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* The patients' age between 7 month and 14 years with a suspected elbow fracture.
* Patients who less than 7 days after the injury of elbow.

Exclusion Criteria:

* Patients with a an open injury in elbow.
* Patients with suspected vascular injury.
* Patients with unstable vital signs .

Ages: 7 Months to 14 Years | Sex: All
Age Groups: Child
Study Population: Ultrasonography examination is done by a 5-10 MHz linear probe. Immediately after it , sonographic fndings are recorded the on data collection forms and after that standard two-view radiographic imaging (AP and lateral elbow X-ray) of the elbow is performed and compared with US results. For performing elbow ultrasonography, patients took a sitting position in front of the examiner. In this position, the elbow flexed to 90 degrees , then the transducer was placed over the posterior-midline aspect of the distal humerus. Both transverse and longitudinal views of the elbow are obtained, and still, pictures and video clips are recorded in each orientation.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2023-08-07 (Estimated); Primary Completion 2024-08-07 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the accuracy of elbow ultrasonography for the diagnosis of elbow fractures in children following trauma. | Base line
  Ultrasonography examination is done by a 5-10 MHz linear probe , searching for fracture sonographic fndings such as fracture line (it's site and size in cm), lipohaemarthrosis, subcutaneous edema, intramuscular haematoma, subperiosteal haematoma and posterior fat pad.
  For performing elbow ultrasonography, patients took a sitting position in front of the examiner. In this position, the elbow flexed to 90 degrees , then the transducer was placed over the posterior-midline aspect of the distal humerus. Both transverse and longitudinal views of the elbow are obtained, and still, pictures and video clips are recorded in each orientation.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Gabeer, Lecturer, Study Director — Assiut University; Hesham Mohammed, Lecturer, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Azizkhani R, Hosseini Yazdi Z, Heydari F. Diagnostic accuracy of ultrasonography for diagnosis of elbow fractures in children. Eur J Trauma Emerg Surg. 2022 Oct;48(5):3777-3784. doi: 10.1007/s00068-021-01648-6. Epub 2021 Mar 24. PMID 33763708